CLINICAL TRIAL: NCT07189182
Title: Clinical Evaluation of the Origin Intubation System
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amit Raj Saxena, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 80068
Record Dates: First submitted 2025-05-30; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Device Usability
Keywords: Intubation; General Anesthesia; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Use of the Origin Intubation System (Experimental): The Origin Intubation System will be utilized on participants undergoing general anesthesia for surgery.
  Interventions: Device: Origin Intubation System

INTERVENTIONS:
Device: Origin Intubation System — This device leverages self-deploying geometry to guide intubation.

SUMMARY:
There are currently two options that are utilized are artificial airways in the operating room as well in emergency medicine: the endotracheal tube and the supraglottic airway. However, with these devices, healthcare professionals often experience difficulty and/or failure in utilizing these devices during their first-pass at intubation. Additionally, military medics often forego intubation in favor of basic life support during prolonged resuscitation. This study aims to test a device, one that has been tested in over 100 cadavers, to determine if it is a viable and safer/more successful option for intubation.

DETAILED DESCRIPTION:
While previous attempts to address the challenge of airway management involve improved visualization tools (still requiring advanced anatomical knowledge), the focus of this clinical study is to evaluate the performance of the Origin Intubation System, which leverages self-deploying geometry to guide intubation. The enabling technology is vine-inspired tip-growth, in which a soft tube extends from its tip into potentially complex shapes, driven only by a low internal air pressure. This paradigm enables a novel device design that aids in intubation through semi-self-navigation, which is resilient to difficult visualization or user skill, is significantly less traumatic compared to existing methods; and fast (because it does not require the user to identify and navigate the internal anatomy).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects 18 years of age or older and less than 75.
2. English or Spanish Speaking.
3. Undergoing elective surgery requiring endotracheal intubation.
4. Use of general anesthesia.

Exclusion Criteria:

1. Patients with high aspiration risk.
2. Inability to provide informed consent in English or Spanish
3. Patients for whom an awake intubation is indicated and planned.
4. Patients with a history of head and neck radiation.
5. Pregnant patients.
6. Patients with BMI >35
7. ASA 4 or higher
8. Patients who the investigator deems ineligible at the investigator's discretion.
9. Planned post-operative intubation.
10. Current incarceration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall intubation duration | Day of surgery.
  The time needed for intubation.

SECONDARY OUTCOMES:
First-pass intubation success | Day of surgery.
  Ability to intubate with the device the first time of use on a given participant.
Overall intubation success | Day of surgery.
  Whether or not the clinician is able to intubate using the Origin Intubation System.
Adverse events | From enrollment to follow-up period.
  Adverse events associated with use of experimental device.
User assessment of intubation | Day of surgery.
  Usability of experimental device.
Patient assessment of intubation | Day of surgery.
  Participant feedback on experimental device, if any.
Patient airway characteristics | Day of surgery.
  Mallampati, thyromental distance, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang HE, Schmicker RH, Daya MR, Stephens SW, Idris AH, Carlson JN, Colella MR, Herren H, Hansen M, Richmond NJ, Puyana JCJ, Aufderheide TP, Gray RE, Gray PC, Verkest M, Owens PC, Brienza AM, Sternig KJ, May SJ, Sopko GR, Weisfeldt ML, Nichol G. Effect of a Strategy of Initial Laryngeal Tube Insertion vs Endotracheal Intubation on 72-Hour Survival in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):769-778. doi: 10.1001/jama.2018.7044. PMID 30167699
- [Background] Karamchandani K, Wheelwright J, Yang AL, Westphal ND, Khanna AK, Myatra SN. Emergency Airway Management Outside the Operating Room: Current Evidence and Management Strategies. Anesth Analg. 2021 Sep 1;133(3):648-662. doi: 10.1213/ANE.0000000000005644. PMID 34153007